CLINICAL TRIAL: NCT06070168
Title: Determining the Effect of Telephone Counseling Service Provided to Primiparous Mothers on Postpartum Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Sümeyye BAL, Ph.D., Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021/485
Record Dates: First submitted 2023-09-30; First posted 2023-10-06 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Depression, Postpartum
MeSH Terms: conditions — Depression, Postpartum | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telephone Counseling (Experimental): Mothers in labor after normal birth at the postpartum clinic At least 6 hours later and for cesarean births, the researcher will visit the patient after 12 hours.
  Mothers will be interviewed according to the inclusion criteria and exclusion criteria, and will be informed about the study.
  will be given and their consent will be taken, the mother information form and the depression form will be filled in, a pre-test will be done and the communication will be completed will get their numbers.
  The researcher will contact the experimental group by phone. He will introduce himself and 6 weeks (during postpartum). It will provide the mother with the consultancy service she needs about herself and the newborn 24 hours a day. After 6 weeks, the training will end and the third researcher will make post-tests of the depression scale to both groups without knowing the experimental and control groups.
  Interventions: Other: Telephone Counseling
- control group (No Intervention)

INTERVENTIONS:
Other: Telephone Counseling — Mothers in labor after normal birth at the postpartum clinic At least 6 hours later and for cesarean births, the researcher will visit the patient after 12 hours.
  Mothers will be interviewed according to the inclusion criteria and exclusion criteria, and will be informed about the study.
  will be given and their consent will be taken, the mother information form and the Edinburgh Postpartum Depression Scale (EPDS) form will be filled in, a pre-test will be done and the communication will be completed.
  will get their numbers. The researcher will contact the experimental group by phone. He will introduce himself and 6 weeks (during postpartum) It will provide the mother with the consultancy service she needs about herself and the newborn 24 hours a day. After 6 weeks, the training will end and the third researcher will make post-tests of the depression scale to both groups without knowing the experimental and control groups.
  Other Names: control group
  Arms: Telephone Counseling

SUMMARY:
The aim of this study is to determine the effect of telephone counseling services provided to primiparous mothers on postpartum depression.

Hypotheses H01; there is no difference between the postpartum depression score of the telephone counseling services group and the postpartum depression score of the control group.

The study will be carried out in two different groups. The practice will start with meeting the women who give birth will be visited by the researcher at the postpartum clinic at least 6 hours after normal birth and 12 hours after cesarean births.

After the women are evaluated in terms of eligibility criteria for the research, the women who are eligible will be informed about the research and written informed consent will be obtained from the women who accept. The random distribution of women to the study groups will be carried out using the Block Randomization method. The following applications will be made to the groups.

The researcher will contact the experimental group by phone. He will introduce herself and 6 weeks (during postpartum). It will provide the mother with the consultancy service she needs about herself and the newborn 24 hours a day. After 6 weeks, the training will end and the third researcher will make post-tests of the depression scale to both groups without knowing the experimental and control groups.

ELIGIBILITY:
Inclusion Criteria:

* primiparous women
* Agreeing to participate in the research and obtaining written permission,
* No hearing or vision problems

Exclusion Criteria:

* multiparous women

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2023-10-07 (Actual); Primary Completion 2024-03-03 (Actual); Study Completion 2024-03-03 (Actual)

PRIMARY OUTCOMES:
Change in postpartum depression | immediately postpartum 6 hours later and immediately after the postpartum 6 weeks later
  Edinburgh Postpartum depression scale Depression Scale

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Ondokuz Mayis University, Samsun, Atakum
  - Ondokuz Mayis University, Samsun

IPD SHARING:
Plan to Share IPD: No